CLINICAL TRIAL: NCT06121570
Title: Phase I Study of Autologous Tumor-Draining Lymph Node-Derived Lymphocytes as Neoadjuvant Therapy for HER2-Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., Director of Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2021] 04-01
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms
Keywords: HER2-Negative; Neoadjuvant Chemotherapy; Lymph Node; Lymphocytes; Adoptive Cell Therapy; Doxorubicin; Epirubicin; Cyclophosphamide; Nab-paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy; Doxorubicin; Epirubicin; Cyclophosphamide; fludarabine; Interleukin-2; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + LNL treatment (Experimental): Participants receive two cycles of doxorubicin or epirubicin, plus cyclophosphamide (AC or EC), followed by neoadjuvant LNL treatment, which consists of non-myeloablative lymphocyte depleting regimen of chemotherapy with cyclophosphamide and fludarabine, followed by infusion of LNL and interleukin-2. After LNL treatment, participants receive four-cycles of nab-paclitaxel as neoadjuvant therapy prior to definitive surgery. The choice of doxorubicin or epirubicin should be the same as the prior neoadjuvant chemotherapy.
  Interventions: Procedure: Sentinel Lymph Node Biopsy (SLNB); Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor-draining lymph node-derived lymphocyte (LNL); Biological: Interleukin-2; Drug: Nab-paclitaxel

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy (SLNB) — A sample of the participant's tumor-draining lymph nodes will be collected and sent to the biotherapy center for LNL isolation and expansion.
  Other Names: SLNB
Drug: Doxorubicin — Doxorubicin will be administered at 60 mg/m^2 IV on Day 1 of Cycles 1-2 of the neoadjuvant chemotherapy of the study.
Drug: Epirubicin — Epirubicin will be administered at 100 mg/m^2 IV on Day 1 of Cycles 1-2 of the neoadjuvant chemotherapy of the study.
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 600 mg/m^2 IV on Day 1 of Cycles 1-2 of the neoadjuvant chemotherapy of the study.
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 500 mg/m^2 IV daily for three days. Cyclophosphamide will be initiated five days prior to the anticipated LNL transfer, and the precise timing will depend on the rate of in vitro LNL growth.
Drug: Fludarabine — Fludarabine will be administered at 30 mg/m^2 IV daily for three days. Fludarabine will be initiated five days prior to the anticipated LNL transfer, and the precise timing will depend on the rate of in vitro LNL growth.
Biological: Tumor-draining lymph node-derived lymphocyte (LNL) — Participants receive single infusion of LNL at the recommended phase 2 dose (RP2D).
  Other Names: LNL
Biological: Interleukin-2 — Eight to twelve hours after completing the LNL infusion, all participants will receive intermediate-dose decrescendo IL-2 IV.
  Other Names: IL-2
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered at 260 mg/m^2 IV on Day 1 of Cycles 3-6 of the neoadjuvant chemotherapy of the study.

SUMMARY:
RATIONALE: Patients with HER2-negative breast cancer not responding to initial neoadjuvant chemotherapy might have lower chances for a pathologic complete response (pCR) at definitive surgery, indicating worse prognosis. Adoptive cell therapy has demonstrated efficacy in advanced breast cancer, but whether the addition of adoptive cell therapy to neoadjuvant chemotherapy could increase the pCR rate remains unclear. Tumor-draining lymph node-derived lymphocytes (LNLs) that have abundant tumor-reactive T cells, but not exhausted T cells, are easy to produce. It is not yet known whether LNL treatment is safe and effective in patients with HER2-negative breast cancer not responding to neoadjuvant chemotherapy.

PURPOSE: This phase I trial is mainly to investigate the safety of autologous LNL in patients with HER2-negative breast cancer not responding to neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the participant must:

1. Have signed the informed consent to study participation.
2. Be a female subject and aged between 18 and 70 years.
3. Provide a core needle biopsy which is histologically confirmed as invasive breast cancer. Excisional biopsy or surgical biopsy is not allowed.
4. Have received two cycles of doxorubicin or epirubicin, plus cyclophosphamide, and had stable disease (SD) confirmed by breast MRI.
5. Have breast cancer defined as the following combined primary tumor (T), regional lymph node (N), and distant metastasis (M) staging per AJCC for breast cancer staging criteria version 8 based on breast MRI assessment before receiving neoadjuvant chemotherapy:

   The minimum size of the primary tumor was 1 cm in largest diameter by breast MRI, N0-3, M0.
6. Have HER2-negative breast cancer, defined as 0-1+ by immunohistochemistry or 2+ by immunohistochemistry without HER2 amplification by FISH.
7. Have known hormone receptor status (estrogen receptor [ER], progesterone receptor [PgR]), Ki67 value and, if institutional standard permits, known tumor grade.
8. Have not received prior therapies for breast cancer, including but not limited to, chemotherapy (except two cycles of doxorubicin or epirubicin, plus cyclophosphamide), radiotherapy, hormonal therapy, targeted therapy, biological therapy, immunotherapy and surgery.
9. Have accessible tumor-draining lymph nodes by surgery to grow LNL. Participants have not received sentinel lymph node biopsy (SLNB) and ipsilateral axillary lymph node dissection (ALND) for the breast cancer lesion.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Demonstrate adequate normal organ function:

    NOTE: Blood component or cytokine therapy is not allowed within 14 days before surgery.
    1. Routine blood test:

       * Absolute neutrophil count (ANC) ≥1.5×10^9/L
       * Lymphocyte count (LC) >0.5×10^9/L
       * Platelets (PLT) ≥100×10^9/L
       * Hemoglobin (Hb) ≥90 g/L
    2. Liver function test:

       * AST and ALT ≤2.5×ULN (≤5×ULN for participants with liver metastases)
       * ALP ≤2.5×ULN (≤5×ULN for participants with liver or bone metastases)
       * Total bilirubin ≤1.5×ULN (≤3.0 mg/dL for participants with Gilbert's syndrome)
    3. Renal function test:

       • Calculated creatinine clearance (CrCL) ≥45 mL/min OR creatinine ≤1.5×ULN
    4. Coagulation function test:

       * APTT ≤1.5×ULN
       * INR or PT ≤1.5×ULN
    5. Doppler echocardiography:

       • Left ventricular ejection fraction (LVEF) ≥50%
    6. Pulmonary function test:

       * FEV1 ≥60%
12. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through one year (or longer as specified by local institutional guidelines) after the last dose of study treatment. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to LNL infusion.
13. Have recovered from prior therapy-related adverse events to Grade≤1 per CTCAE version 5.0 criteria or met the criteria of normal organ function specified above prior to the surgery for obtaining the lymph nodes, except for second-degree peripheral nerve injury, alopecia, leukoderma, hypothyroidism controlled by thyroid hormone replacement therapy, type 1 diabetes controlled by insulin therapy, and other irreversible toxic events that would not be exacerbated by LNL infusion as judged by the investigator (e.g., hearing loss).

Exclusion Criteria:

The participant must be excluded from participating in this trial if the participant:

1. Has metastatic breast cancer.
2. Has a known additional malignancy that is progressing or requires active treatment within the last 5 years. Exceptions include basal or squamous cell carcinoma of the skin, and thyroid cancer that has undergone potentially curative therapy or in situ cervical cancer.
3. Has a known history of cardiovascular disease, including but not limited to, (1) congestive heart failure (New York Heart Association [NYHA] functional classification Class > 2), (2) unstable angina pectoris, (3) myocardial infarction in the past 3 months, (4) supraventricular arrhythmia or ventricular arrhythmia that requires treatments.
4. Has interstitial pneumonia or active pneumonia that has clinical implications, or other respiratory diseases that seriously affect pulmonary function.
5. Has an active infection requiring systemic therapy or has an unexplained fever of >38.5℃ except fevers caused by cancer.
6. Has arterial and/or venous thrombotic events in the past 5 months, e.g., cerebrovascular accident, deep vein thrombosis or pulmonary embolism.
7. Has a known psychiatric, alcohol abuse or substance abuse disorders.
8. Is pregnant or breastfeeding.
9. Has an active autoimmune disease, a history of autoimmune disease, or autoimmune disease that has required systemic treatment (e.g., with use of prednisone at a dose of >10 mg per day or other corticosteroids at an equivalent dose). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
10. Has a history of congenital immunodeficiency or acquired immunodeficiency (e.g., positive serology test for HIV).
11. Has tuberculosis in the past one year, or has a history of active tuberculosis more than one year but did not receive regular treatments.
12. Has known active hepatitis B or hepatitis C. Participants that are hepatitis B surface antigen (HBsAg) or hepatitis B core antigen (HBcAg) positive may participate provided that the HBV DNA level is normal. Participants that are hepatitis C antibody positive may participate provided that the HCV DNA level is normal. Carriers of HBV or HCV must receive anti-virus therapy, and take regular DNA copy number tests during this trial.
13. Has received a live vaccine within 4 weeks prior to enrollment, or plans to receive a live vaccine during this trial.
14. Has a history of allogeneic bone marrow or organ transplant.
15. Has received the study-related drugs including anthracycline, cyclophosphamide, taxane, fludarabine, interleukin-2, except two-cycle neoadjuvant chemotherapy of doxorubicin or epirubicin, plus cyclophosphamide.
16. Has a history of hypersensitivity or allergy to the drugs in this study and any of their components including but not limited to, LNL, doxorubicin/epirubicin, cyclophosphamide, nab-paclitaxel, fludarabine, interleukin-2, dimethyl sulphoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (β-lactam antibiotics, gentamicin).
17. Has contraindication for use of IL-2, including but not limited to, refractory or intractable epilepsy, and active gastrointestinal bleeding.
18. Has a history of Grade≥2 neuropathy.
19. Has received long half-life angiogenesis inhibitors within four weeks prior to enrollment, e.g., bevacizumab.
20. Is receiving any medication prohibited in combination with study treatments as described in the respective product labels, unless medication was stopped within 7 days prior to enrollment.
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with participation for the full duration of the study, or render study participation not compatible with the participant's best interest, in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | From the LNL infusion up to 28 days post-infusion
  Adverse events are reported based upon Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. DLT will be defined as a non-hematologic Grade 3 or higher adverse event, occurring within the 28 days immediately after LNL infusion, that is probably or definitely related to LNL infusion, and lasts more than 28 days or does not resolve to Grade<3 despite treatment with dexamethasone at 10 mg per 12 hours IV for 7 days (or other corticosteroid at equivalent dose), and/or tocilizumab at 8mg/kg IV for three times.
Incidence of Grade≥3 Treatment-Emergent Adverse Event (TEAE) | From the LNL infusion up to 28 days post-infusion
  Adverse events are reported based upon CTCAE version 5.0 criteria. The incidence of Grade≥3 TEAE occurring within the 28 days immediately after LNL infusion will be summarized with descriptive statistics.

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 at the time of definitive surgery | Up to approximately 26~29 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy assessed by the local pathologist at the time of definitive surgery.
Objective Response Rate (ORR) | Up to approximately 26~29 weeks
  Objective response rate is defined as the percentage of participants in the analysis population who have achieved complete response (CR) or partial response (PR) assessed by modified RECIST criteria by breast MRI during the study. The percentage of participants who experienced a CR or PR is presented.
6-month, 1-year and 2-year Event-Free Survival (EFS) | Up to approximately two years
  Event-free survival is defined as the time from enrollment to the first date of disease progression while on primary therapy or disease recurrence (local, regional, distant, invasive contralateral breast) after surgery or death due to any cause. Patients who terminate the study without evidence of any of the above events will be censored at the date of their last follow-up tumor assessment. Patients who start a new anti-tumor therapy (with the exception of adjuvant endocrine therapy in ER or PgR positive tumors after surgery) in the absence of disease progression or recurrence will be censored at their last follow-up tumor assessment before the start of the new therapy.
Overall Survival (OS) | Up to approximately five years
  Overall survival is defined as the time from enrollment to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Levels of multiple different cytokines in blood samples before and after LNL infusion. | Up to approximately two years
  Levels of multiple different cytokines in blood samples including Granzyme B, IFN-γ, GM-CSF, IL-2, IL-4, IL-6, etc. will be measured using cytokine chips, ELISA or flow cytometry at various time points before and after LNL infusion.
Distribution of T cell subsets in blood samples before and after LNL infusion. | Up to approximately two years
  Distribution of T cell subsets in blood samples will be measured using flow cytometry at various time points before and after LNL infusion.
Distribution of T-cell receptor (TCR) clonotype in blood samples before and after LNL infusion. | Up to approximately two years
  Distribution of T-cell receptor (TCR) clonotype in blood samples will be measured using TCR sequencing at various time points before and after LNL infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, M.D., Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China